CLINICAL TRIAL: NCT05897242
Title: ACT on Vaping: Digital Therapeutic for Young Adult Vaping Cessation
Brief Title: A Smartphone Application (ACT on Vaping) for Vaping Cessation in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jaimee Heffner, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG1122763; NCI-2022-10010 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UG3DA057032 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Nicotine Dependence; Nicotine Addiction; Nicotine Use Disorder; Nicotine Vaping; Vaping
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Any outcome evaluator who has direct contact with participants will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Act on Vaping app) (Experimental): Participants receive supportive messages and use the ACT on Vaping smartphone app. They also receive incentivized text message check-ins assessing their vaping status.
  Interventions: Behavioral: Smartphone app; Other: Text Message; Other: Survey Administration
- Arm II (Incentivized text message check-ins) (Active Comparator): Participants receive incentivized text messages check-ins assessing their vaping status.
  Interventions: Other: Text Message; Other: Survey Administration

INTERVENTIONS:
Behavioral: Smartphone app — Use ACT on Vaping smartphone app
  Other Names: ACT on Vaping
  Arms: Arm I (Act on Vaping app)
Other: Text Message — Receive text messages
  Other Names: SMS Text
Other: Survey Administration — Ancillary studies

SUMMARY:
Almost one in ten young adults report current e-cigarette use, putting them at risk of developing nicotine addiction and long-term health effects of exposure to inhaled toxicants. Despite the need for effective treatments to help these young users quit, very few treatments targeting any type of tobacco use among young adults have been evaluated, particularly for young adults who vape and have unique treatment needs. To address these needs, this trial will evaluate a digital program for young adult e-cigarette users at all stages of readiness to quit called ACT on Vaping.

DETAILED DESCRIPTION:
OUTLINE:

Participants are randomized to 1 of 2 arms.

ARM I: Participants use the ACT on Vaping smartphone app and text messaging program and receive incentivized text messages assessing their vaping status.

ARM II: Participants receive incentivized text messages check-ins assessing their vaping status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30.
* Current weekly user of e-cigarette product(s).
* Owns an Android phone or iPhone.
* Has an email address.
* United States (US) resident, with a US mailing address.
* Willing to complete all study procedures.

Exclusion Criteria:

* Currently using other tobacco cessation treatments at the time of screening, including pharmacotherapy or behavioral support (note: use of these treatments is allowable during trial participation).
* Member of the same household as another research participant.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via the Facebook/Instagram advertising platform. Two hundred individuals were eligible. The final sample comprised 61 participants who were randomized in January 2024.
Period: Overall Study
Arm/Group | Arm I (Act on Vaping App) | Arm II (Incentivized Text Message Check-ins)
Started | 31 | 30
Completed | 23 | 29
Not Completed | 8 | 1
Not completed — Lost to Follow-up | 6 | 1
Not completed — Incomplete | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Act on Vaping App) | Arm II (Incentivized Text Message Check-ins) | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (3.2) | 22 (3.6) | 21.8 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 9 | 17 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 27 | 49
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Vaping frequency (past 30 days) [Count of Participants; unit: Participants]
  Once a week or more but not daily | 6 | 0 | 6
  At least daily | 25 | 30 | 55
Vaping intensity (past 30 days) [Count of Participants; unit: Participants]
  0-4 times/day | 6 | 1 | 7
  5-9 times/day | 10 | 7 | 17
  10-14 times/day | 4 | 6 | 10
  15-19 times/day | 5 | 5 | 10
  20-29 times/day | 3 | 5 | 8
  30+ times/day | 3 | 6 | 9
Other tobacco product use (past 30 days) [Count of Participants; unit: Participants]
  Not at all | 15 | 13 | 28
  Less than once a month | 5 | 8 | 13
  Once a month or more, but less than once a week | 4 | 3 | 7
  Once a week or more, but not daily | 4 | 2 | 6
  At least daily | 3 | 4 | 7
24-hour quit attempts (past 12 months) [Count of Participants; unit: Participants]
  At least 1 attempt | 26 | 21 | 47
  No attempts | 5 | 9 | 14
Contemplation Ladder Score [Count of Participants; unit: Participants]
  High quit readiness (>5) | 24 | 24 | 48
  Low quit readiness (≤ 5) | 7 | 6 | 13
e-cigarette Fagerström Test for Nicotine Dependence (e-FTND) [Mean (Standard Deviation); unit: units on a scale] — Range of scores is 0-10. Higher values represent greater severity of dependence.
  units on a scale | 5 (2.2) | 5.4 (2.5) | 5.2 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Overall Treatment Satisfaction Rating
Description: We calculated descriptive statistics (mean, standard deviation) for the primary acceptability benchmark of overall satisfaction averaging at least 3.5 on a 1-5 Likert-type scale within the ACT on Vaping arm only.
  Overall satisfaction was assessed with a 5-point Likert-type item on the 3-month follow-up survey, with response options ranging from (1) "not at all" to (5) "very much." The ACT on Vaping benchmark average of 3.5 falls between ratings of 3="somewhat" and 4="mostly." Higher values are associated with a higher level of satisfaction.
Time Frame: At 3 months post-randomization
Population: We calculated descriptive statistics (e.g., means, proportions) for the ACT on Vaping treatment group to evaluate the go/no-go criteria and to compare the two arms on other indicators of treatment acceptability and efficacy. Given that pilot and feasibility trials are not appropriate designs for testing hypotheses regarding the efficacy of interventions, we focused on descriptive differences as an alternative to hypothesis testing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Act on Vaping App)
Number analyzed (Participants) | 21
units on a scale | 3.8 (1.3)

2. Primary Outcome: Change in Readiness to Quit
Description: Will evaluate differences of Contemplation Ladder scores. The 1-item Contemplation Ladder, scores range from 0-10, was used to assess readiness to quit using e-cigarettes. The higher the score, the more ready the person is to make a change. The anchor for the cut-off score of 5, indicating high vs. low quit readiness, is "Think I should quit but not quite ready."
Time Frame: From baseline to 3 months post-randomization
Population: We calculated descriptive statistics (e.g., means, proportions) for the ACT on Vaping treatment group to evaluate the go/no-go criteria and to compare the two arms on other indicators of treatment acceptability and efficacy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Act on Vaping App) | Arm II (Incentivized Text Message Check-ins)
Number analyzed (Participants) | 24 | 29
units on a scale | 0.96 (2.0) | 0.72 (1.7)

3. Primary Outcome: Percentage of Participants With a 24-hour Quit Attempt
Description: Making a 24-hour quit attempt between baseline and 3-month follow-up was assessed via self-report at the 3-month follow-up survey. The percentage of participants with self-reported 24-hour quit attempts is evaluated descriptively.
Time Frame: At 3 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Act on Vaping App) | Arm II (Incentivized Text Message Check-ins)
Number analyzed (Participants) | 24 | 29
Participants | 21 | 22

4. Primary Outcome: Cotinine-confirmed 30-day Point Prevalence Abstinence From All Nicotine and Tobacco
Description: Complete case, self-reported 30-day abstinence from all nicotine and tobacco products at 3 months, confirmed via saliva cotinine testing. Differences were evaluated descriptively.
Time Frame: At 3 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Act on Vaping App) | Arm II (Incentivized Text Message Check-ins)
Number analyzed (Participants) | 24 | 29
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected by a web-based survey (on Day 21, 42, 63, and at the 3-month follow-up time point).
Description: Adverse events were collected by a web-based survey, and their relationship to the intervention was adjudicated by an independent medical monitor.
Arm/Group | Arm I (Act on Vaping App) | Arm II (Incentivized Text Message Check-ins)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 1/31 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Act on Vaping App) (N=31) | Arm II (Incentivized Text Message Check-ins) (N=30)
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — The lingering symptoms of COVID- 19 may be influenced by the trial.
Worsening of pre-existing mental health condition (Psychiatric disorders) | 0 (0) | 1 (1) — Worsening of a pre-existing mental health condition.
Lowered resting heart rate (Cardiac disorders) | 1 (1) | 0 (0) — The participant reported an extremely lowered resting heart rate of 45 BPM after quitting smoking a few days prior.
Burn on inner thigh. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Burn to inner thigh from laptop battery.

LIMITATIONS AND CAVEATS:
A limitation of this study is the small sample size, which, while appropriate for a pilot study, does not allow for a definitive evaluation of acceptability or efficacy and limits the generalizability of the findings. Additionally, the cotinine testing for biochemical verification of abstinence was not directly observed, leaving open the possibility that the test could have been completed by someone other than the participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT05897242/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT05897242/ICF_000.pdf